CLINICAL TRIAL: NCT05293366
Title: LOng COvid COmorbidities: Evaluation of Endocrine, Metabolic, Neuropsychiatric, Muscle, Cardiovascular, Pulmonary and Dermatologic Functions
Brief Title: LOng COvid COmorbidities: Endocrine,Metabolic,Neuropsychiatric,Muscle,Cardiovascular,Pulmonary,Dermatologic Dysfunctions
Acronym: LO-COCO
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Annamaria Colao, Clinical Professor, Federico II University
Other Study IDs: LO-COCO
Record Dates: First submitted 2022-03-19; First posted 2022-03-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Long Covid-19
Keywords: Long Covid-19; Endocrine Complications; Metabolic Complications; Neuropsychiatric Complications; Muscular Complications; Cardiovascular Complications; Pulmonary Complications; Dermatologic Complications
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessments of endocrinological phenotypes of LO-COCO patients — Assessment of:thyroid-stimulating hormone(TSH),free triiodothyronine (FT3), free thyroxine (FT4),calcitonin,antibodies against thyroglobulin (AbTG) and against thyroperoxidase (AbTPO),adrenocorticotropic hormone (ACTH),cortisol, luteinizing hormone (LH),follicle-stimulating hormone(FSH),Testosterone,17-beta estradiol,sex hormone binding globulin (SHBG),progesterone, prolactin (PRL), growth hormone (GH), insulin growth factor-1 (IGF-1), dehydroepiandrosterone sulphate (DHEAS),delta 4-androstenedione,aldosterone,renin,glycemia, insulinemia, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, HbA1c, vitamin D, adiponectin, irisin, IL-6.Thyroid and ovarian ultrasounds, pituitary and adrenal MRI will be performed as well. Body composition will be assessed with bioimpedance analysis and DXA scans.Female sexual dysfunctions will be evaluated with Female Sexual Function Index (FSFI), Sexual Inhibition and Sexual Excitation Scale (SIS/SES),Body Uneasiness Test (BUT).
  Other Names: Evaluation of hormonal and metabolic health
Diagnostic Test: Assessment of muscular phenotypes of LO-COCO patients — Questions will be collected regarding the tolerance to physical activity and modifications after diagnosis of Covid. Muscular strength will be assessed by means of tests (Medical Research Council Scale) and dynamometers. Balance will be assessed with a Romberg test, tolerance to stress will be assessed by means of cyclometer.
Diagnostic Test: Assessment of neuropsychiatric phenotypes of LO-COCO patients — Validated questionnaires will be collected to investigate depression (Beck Depression Inventory-II, BDI-II), apathy (Apathy Evaluation Scale, AES), anxiety (Test Anxiety Inventory, TAI), attention and cognitive functions (Montreal Cognitive Assessment and Quick Mild Cognitive Impairment). Fatigue will be assessed by Fatigue Rating Scale (FRS) and Fatigue Severity Scale (FSS). Muscle power will be assessed by six-minute walking test and sit and stand up test. The presence of myopathy will be evaluated by mean electrophysiological study.
Procedure: Muscle biopsy — Muscle biopsy will be performed upon need.
Diagnostic Test: Assessment of pulmonary phenotypes of LO-COCO patients — Modified Medical Research council questionnaire will be administered for evaluating of the dyspnoea level. Complete respiratory status assessment, including global spirometry, CO lung diffusion capacity and arterial gases analysis will be run. HRCT - high resolution CT scan of the chest - will be performed in selected cases to rule out the eventual sequelae of SARS-Cov2 related pneumonia.
Diagnostic Test: Assessment of cardiological phenotypes of LO-COCO patients — Cardiological assessment will be run upon data collected from: Short Form-36 Health Survey (SF36), echocardiogram at rest and during stress tests, six-minute walking test, N-terminal fragment brain natriuretic peptides (NT-proBNP)
Diagnostic Test: Assessment of vascular phenotypes of LO-COCO patients — The assessment of the potential post-thrombotic vascular damage will comprise the investigation of prevalence of previously unknown deep venous thrombosis by ultrasonography.
Diagnostic Test: Assessment of dermatological phenotypes of LO-COCO patients — Dermatology evaluation will account on: thrichoscopy, dermoscopy, onychoscopy and capillaroscopy, confocal microscopy, skin ultrasonography
Procedure: Tissue biopsy — Tissue biopsy will be performed upon need.

SUMMARY:
Considering the compelling amount of studies focused on patients in the active phase of COVID-19 disease and the scarcity of studies focused on patient cured from disease aimed at evaluating the sequelae of SARS-CoV-2 infection, the purpose of the study is to investigate whether in patients recovered from COVID-19 disease, SARS-CoV-2 infection has induced: 1) endocrine-metabolic function damage; 2) neuro-psychiatric damage; 3) muscle damage; 4) pulmonary damage; 5) cardiological damage; 6) venous vascular damage; 7) dermatological damage. Patients will be evaluated at baseline (at discharge from infectious and/or pneumology unit) and after 3- 12 months. A better definition of the prevalence and type of sequelae after recovery from COVID-19 disease could significantly improve the therapeutic management and long-term follow-up of these patients, with a relevant impact in terms of health resources and public health.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether in patients recovered from COVID-19 disease, SARS-CoV-2 infection has induced: 1) Endocrine-metabolic function damage, 2) Neuro-psychiatric damage, 3) Muscle damage, 4) Pulmonary damage, 5) Cardiological damage, 6) Post-thrombotic vascular damage, 7) Dermatological damage.

The assessment of the potential endocrine-metabolic function damage will comprise the investigation of alterations in particular in: thyrotropic axis (prevalence of hypothyroidism and alterations of the thyroid gland); female gonadotropic axis (prevalence of hypogonadism) with assessment of potentially impaired reproductive and sexual function (prevalence of morpho-structural alterations of the ovary, sexual dysfunction); corticotropic axis (prevalence of hypoadrenalism and alterations of the adrenal gland); somatotropic axis (prevalence of growth hormone deficiency); lactotropic axis (prevalence of hyperprolactinaemia); metabolic profile (prevalence of metabolic syndrome, overweight, obesity, insulin resistance, type 2 diabetes mellitus, dyslipidemia, hypovitaminosis D).

The assessment of the potential neuro-psychiatric damage will comprise the investigation of prevalence of depression, alteration in the quality of life, apathy, anxiety, deficit of attention and cognitive skills.

The assessment of the potential muscle damage will comprise the investigation of prevalence of fatigue, reduced resistance and muscle strength, reduced muscle power, reduced exercise tolerance, myopathy.

The assessment of the potential pulmonary damage will comprise the investigation of prevalence of parenchymal sequelae of interstitial/organized pneumonia, lung dysfunctions, dyspnoea.

The assessment of the potential cardiological damage will comprise the investigation of prevalence of echocardiographic changes at rest and during echocardiogram stress tests, dysfunctions in cardiopulmonary performance.

The assessment of the potential post-thrombotic vascular damage will comprise the investigation of prevalence of previously unknown deep venous thrombosis.

The assessment of the potential dermatological damage will comprise the investigation of prevalence of cutaneous and mucosal lesions, defluvium with identification of specific trichoscopic patterns and onychopathies with identification of specific onychoscopic/capillaroscopic patterns.

Patients will be evaluated at baseline (at discharge from infectious and/or pneumology unit) and after 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes recovered from SARS-CoV-2 infection (two negative nasopharyngeal swabs, negative IgM and positive anti SARS-CoV-2 IgG);
* Aged over 18 years of age;
* Ability to understand protocol procedures

Exclusion Criteria:

* Any psychological/psychiatric/other medical conditions compromising the understanding of the nature and purpose of the study, and of its possible consequences
* uncooperative attitude of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients of both sexes recovered from SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Identification of the most frequent phenotypes of Long-COVID syndrome among for COVID-19 patients recently hospitalized and dismissed | Change from baseline at 3-12 months
  This pilot study will allow identifying the frequency and type of endocrinologic, muscular, cardiovascular, pulmonary, dermatological, metabolic and neuropsychiatric disorders that contribute to the long covid syndrome .

SECONDARY OUTCOMES:
Thyroid dysfunctions | Change from baseline at 3-12 months
  Prevalence of thyroid dysfunctions (hypo, hyper functions; thyroiditis)
Female gonadal dysfunctions | Change from baseline at 3-12 months
  Prevalence of female gonadal dysfunctions (hypogonadism and female sexual dysfunctions)
Adrenal dysfunctions | Change from baseline at 3-12 months
  Prevalence of adrenal dysfunctions (hypocortisolism)
Pituitary dysfunctions | Change from baseline at 3-12 months
  Prevalence of pituitary dysfunctions (hyperprolactinemia, GH deficiency)
Metabolic dysfunctions | Change from baseline at 3-12 months
  Prevalence of metabolic dysfunctions (metabolic syndrome, type 2 diabetes, overweight, obesity, insulin-resistance, dyslipidemia, hypovitaminosis D)
Neuro-psychiatric dysfunctions | Change from baseline at 3-12 months
  Prevalence of depression, alteration of the quality of life, apathy, anxiety, deficit of attentional and cognitive skills
Muscle dysfunctions | Change from baseline at 3-12 months
  Prevalence of fatigue, reduced resistance and muscle strength, reduced muscle power, reduced exercise tolerance, myopathy.
Pulmonary dysfunctions | Change from baseline at 3-12 months
  Prevalence of persisting respiratory discomfort in relation to lung function and radiological outcomes (interstitial/organized pneumonia, pulmonary fibrosis)
Cardiological dysfunctions | Change from baseline at 3-12 months
  Prevalence of echocardiographic changes at rest and during echocardiogram stress tests, dysfunctions in cardiopulmonary performance
Post-thrombotic vascular dysfunctions | Change from baseline at 3-12 months
  Prevalence of previously unknown deep venous thrombosis
Dermatological dysfunctions | Change from baseline at 3-12 months
  Prevalence of cutaneous and mucosal lesions, defluvium with identification of specific trichoscopic patterns and onychopathies with identification of specific onychoscopic/capillaroscopic patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, Prof, Principal Investigator — Federico II University
Locations (1):
- Federico II University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auriemma RS, Pirchio R, Liccardi A, Scairati R, Del Vecchio G, Pivonello R, Colao A. Metabolic syndrome in the era of COVID-19 outbreak: impact of lockdown on cardiometabolic health. J Endocrinol Invest. 2021 Dec;44(12):2845-2847. doi: 10.1007/s40618-021-01563-y. Epub 2021 May 26. PMID 34037973
- [Background] Fabbrocini G, Vastarella M, Nappa P, Annunziata MC, Camela E, Greco V, Gaudiello F, Alessio M, Pierri L, Catzola A, Guarino A. A new dermoscopic pattern for chilblain-COVID-19-like skin lesions in adolescents. JAAD Case Rep. 2020 Dec;6(12):1271-1274. doi: 10.1016/j.jdcr.2020.09.024. Epub 2020 Oct 1. No abstract available. PMID 33020736
- [Background] Ortelli P, Ferrazzoli D, Sebastianelli L, Engl M, Romanello R, Nardone R, Bonini I, Koch G, Saltuari L, Quartarone A, Oliviero A, Kofler M, Versace V. Neuropsychological and neurophysiological correlates of fatigue in post-acute patients with neurological manifestations of COVID-19: Insights into a challenging symptom. J Neurol Sci. 2021 Jan 15;420:117271. doi: 10.1016/j.jns.2020.117271. Epub 2020 Dec 14. PMID 33359928
- [Background] Ocampo-Garza SS, Vastarella M, Nappa P, Cantelli M, Fabbrocini G. Telogen effluvium in the new SARS-CoV-2 era. Int J Dermatol. 2021 Jul;60(7):e265-e266. doi: 10.1111/ijd.15482. Epub 2021 Mar 4. No abstract available. PMID 33660272
- [Background] Pivonello R, Auriemma RS, Pivonello C, Isidori AM, Corona G, Colao A, Millar RP. Sex Disparities in COVID-19 Severity and Outcome: Are Men Weaker or Women Stronger? Neuroendocrinology. 2021;111(11):1066-1085. doi: 10.1159/000513346. Epub 2020 Nov 26. PMID 33242856
- [Background] Muscogiuri G, Barrea L, Savastano S, Colao A. Nutritional recommendations for CoVID-19 quarantine. Eur J Clin Nutr. 2020 Jun;74(6):850-851. doi: 10.1038/s41430-020-0635-2. Epub 2020 Apr 14. No abstract available. PMID 32286533
- [Background] Muscogiuri G, Pugliese G, Barrea L, Savastano S, Colao A. Commentary: Obesity: The "Achilles heel" for COVID-19? Metabolism. 2020 Jul;108:154251. doi: 10.1016/j.metabol.2020.154251. Epub 2020 Apr 27. No abstract available. PMID 32353356
- [Background] Isidori AM, Arnaldi G, Boscaro M, Falorni A, Giordano C, Giordano R, Pivonello R, Pofi R, Hasenmajer V, Venneri MA, Sbardella E, Simeoli C, Scaroni C, Lenzi A. COVID-19 infection and glucocorticoids: update from the Italian Society of Endocrinology Expert Opinion on steroid replacement in adrenal insufficiency. J Endocrinol Invest. 2020 Aug;43(8):1141-1147. doi: 10.1007/s40618-020-01266-w. Epub 2020 Apr 25. No abstract available. PMID 32335855
- [Background] Bellastella G, Maiorino MI, Esposito K. Endocrine complications of COVID-19: what happens to the thyroid and adrenal glands? J Endocrinol Invest. 2020 Aug;43(8):1169-1170. doi: 10.1007/s40618-020-01311-8. Epub 2020 Jun 1. No abstract available. PMID 32488724
- [Background] Agarwal S, Agarwal SK. Endocrine changes in SARS-CoV-2 patients and lessons from SARS-CoV. Postgrad Med J. 2020 Jul;96(1137):412-416. doi: 10.1136/postgradmedj-2020-137934. Epub 2020 Jun 11. PMID 32527756
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] D'Alto M, Marra AM, Severino S, Salzano A, Romeo E, De Rosa R, Stagnaro FM, Pagnano G, Verde R, Murino P, Farro A, Ciccarelli G, Vargas M, Fiorentino G, Servillo G, Gentile I, Corcione A, Cittadini A, Naeije R, Golino P. Right ventricular-arterial uncoupling independently predicts survival in COVID-19 ARDS. Crit Care. 2020 Nov 30;24(1):670. doi: 10.1186/s13054-020-03385-5. PMID 33256813
- [Background] Evans PC, Rainger GE, Mason JC, Guzik TJ, Osto E, Stamataki Z, Neil D, Hoefer IE, Fragiadaki M, Waltenberger J, Weber C, Bochaton-Piallat ML, Back M. Endothelial dysfunction in COVID-19: a position paper of the ESC Working Group for Atherosclerosis and Vascular Biology, and the ESC Council of Basic Cardiovascular Science. Cardiovasc Res. 2020 Dec 1;116(14):2177-2184. doi: 10.1093/cvr/cvaa230. PMID 32750108